CLINICAL TRIAL: NCT05874908
Title: Identifying the Microorganisms Responsible for Acute Head and Neck Infections.
Brief Title: Microbiology Studies of Acute Head and Neck Infections
Status: Enrolling by invitation | Type: Observational
Sponsor: The University of Northampton (Other)
Collaborators: Northampton General Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Jazmine Cox, Principal Investigator, The University of Northampton
Other Study IDs: UNorthampton FAST PhD
Record Dates: First submitted 2023-05-08; First posted 2023-05-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial isolates from pus swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Acute head and neck infections cause significant pain and discomfort for patients and impact on their quality of life. Effective antibiotic and surgical treatments have been developed for these infections but they are still able to develop into life-threatening diseases such as meningitis and sepsis. The direct cause of acute head and neck infections is often unknown but it has been suggested that they are due to a disturbance of the normal bacterial growing in the mouth or are from dental origin.

The most common microorganisms identified from these infections in published studies are a group of bacteria known as viridans group streptococci (VGS). There are over 30 individual species of bacteria in the viridans group and VGS are difficult to identify to the level of a single species because of their variability. There is a lack of species identification within the hospital setting and this project aims to gain a deeper understanding of the microorganisms causing acute head and neck infections, focusing on identification of individual species of VGS bacteria.

The investigators will analyse bacterial DNA to determine which species have been identified and will also look at patient data and clinical outcomes (eg. length of hospital stay) to determine if the species causing the infection has any effect on patients.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Suffering with acute head and neck infection of Streptococci.
* Samples must come from Northampton General Hospital.
* Consent to participate in research with at least 24 hours of consideration.

Exclusion Criteria:

* Age <18 years.
* Samples from other National Health Service (NHS) hospitals.
* Infections from other areas of the body.
* Infection identified as caused by non-streptococcal bacteria.
* Chosen not to participate in research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute head and neck infections at Northampton General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2026-04-19 (Estimated); Study Completion 2026-04-19 (Estimated)

PRIMARY OUTCOMES:
Identification of Streptococci Species | 4 years
  Identification by DNA analysis of ribosomal ribonucleic acid (rRNA) genes and biochemical testing.

SECONDARY OUTCOMES:
Patient Characteristics | 4 Years
  Age in years. All measurements will be combined to determine common traits in acute head and neck infections.
Patient Characteristics | 4 Years
  Sex as biological gender. All measurements will be combined to determine common traits in acute head and neck infections.
Patient Characteristics | 4 Years
  Site of Infection in areas of the head and neck. All measurements will be combined to determine common traits in acute head and neck infections.
Clinical Outcomes | 4 Years
  Length of hospital stay in days. All measurements will be combined to determine common traits in acute head and neck infections.
Clinical Outcomes | 4 Years
  Antibiotic treatment in medication type. All measurements will be combined to determine common traits in acute head and neck infections.
Clinical Outcomes | 4 Years
  Diabetic diagnosis in diabetic/non-diabetic. All measurements will be combined to determine common traits in acute head and neck infections.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Woodacre, PhD, BSc, Principal Investigator — University of Northampton
Locations (1):
- University of Northampton, Northampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only share pseudonymised data of participant/clinical outcomes.
Supporting Information: Study Protocol
Time Frame: October 2025
URL: http://pure.northampton.ac.uk/en/impacts/identification-of-the-microorganisms-responsible-for-acute-head-a

REFERENCES:
- See also: Access to dataset, results summary, Doctor of Philosophy (PhD) thesis, publications and impact. — http://pure.northampton.ac.uk/en/impacts/identification-of-the-microorganisms-responsible-for-acute-head-a